CLINICAL TRIAL: NCT04900883
Title: Nurse Perspectives Regarding Use of the Labor Mirror
Status: Completed | Type: Observational
Sponsor: Mount Carmel Health System (Other)
Responsible Party: Principal Investigator, Robin Driver, Perinatal Research Nurse, Mount Carmel Health System
Other Study IDs: 210504-1
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Second Stage Labor
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey — anonymous survey

SUMMARY:
The objective of the study is to examine the views of Labor & Delivery nurses regarding use of the labor mirror during the active phase of the second stage of labor.

DETAILED DESCRIPTION:
A survey link will be sent to Labor & delivery nurses via hospital group email. The nurses will be asked to share their experiences regarding the following: if use of the labor mirror helps patients push more effectively, how often patients accept the labor mirror, why they feel patients may decline use of the labor mirror, how often they offer the labor mirror to eligible patients, and a range of how long they have been a labor & delivery nurse at this facility. The survey is voluntary and the results are anonymous.

ELIGIBILITY:
Inclusion Criteria:

* Labor & Delivery Nurses at Mount Carmel East Hospital

Exclusion Criteria:

* All others

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Labor & Delivery Nurses who work at Mount Carmel East Hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
L&D Nurse views regarding use of the labor mirror | survey will be open for one month
  Does use of the labor mirror help patients push more effectively?

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Carmel Health System, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
The survey is anonymous, so individual results are unknown. However, I do plan to share group results.